CLINICAL TRIAL: NCT06740201
Title: A Clinical Validation Study to Evaluate the Accuracy of a Target Controlled Infusion Model of Cipepofol in Patients With General Anesthesia During Elective Surgery
Brief Title: A Study to Evaluate the Accuracy of aTCI Model of Cipepofol in Patients With General Anesthesia During Elective Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSK3486-408
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cp=0.9μg/ml (Experimental): Plasma target-controlled concentration 0.9μg/ml
  Interventions: Drug: Cipepofol
- Cp=1.2μg/ml (Experimental): Plasma target-controlled concentration 1.2μg/ml
  Interventions: Drug: Cipepofol

INTERVENTIONS:
Drug: Cipepofol — Adjust plasma target-controlled concentration
  Other Names: HSK3486

SUMMARY:
This study is a multi-center (each center independently conducts the study according to the same research protocol), randomized, and open-label clinical study. The main objective is to verify and optimize the accuracy of the target-controlled infusion model of cipepofol.

DETAILED DESCRIPTION:
Subjects who meet the enrollment criteria will be randomly assigned at a 1:1 ratio to two groups with different plasma target-controlled concentrations (Cp) during the induction period: the low-concentration group (Group L) with a concentration of 0.9 μg/ml and the high-concentration group (Group H) with a concentration of 1.2 μg/ml. An interim analysis will be conducted after approximately 5% of the subject data has been collected in each group, including but not limited to indicators such as the effect-site equilibrium rate constant (Ke0).

ELIGIBILITY:
Inclusion Criteria:

* Inpatient patients scheduled for elective surgeries that require tracheal intubation under general anesthesia, with the expected duration of surgery being ≥ 1 hour, excluding those in emergency, cardiothoracic, or neurosurgery departments (patients whose planned surgical types may affect the collection of the Bispectral Index (BIS) are not eligible for enrollment).
* Either male or female, aged ≥ 18 and ≤ 65 years old.
* Classified as grade I - III by the American Society of Anesthesiologists (ASA).
* Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m².
* Vital signs during the screening period meet the following criteria:

Respiratory rate ≥ 10 and ≤ 24 breaths per minute. Pulse oxygen saturation (SpO2) ≥ 95% when breathing air. Systolic blood pressure (SBP) ≥ 90 mmHg and ≤ 160 mmHg. Diastolic blood pressure (DBP) ≥ 60 mmHg and ≤ 100 mmHg. Heart rate ≥ 55 and ≤ 100 beats per minute. (Note: The heart rate result of the 12-lead electrocardiogram (12-ECG) examination after signing the Informed Consent Form (ICF) shall be used as the basis for judgment.)

● Able to understand the procedures and methods of this study, willing to sign the informed consent form and strictly comply with the trial protocol to complete this study.

Exclusion Criteria:

* Those with contraindications for general anesthesia or a history of previous anesthesia accidents.
* Those known to be allergic to the excipients of cipepofol injection (soybean oil, glycerol, triglycerides, egg yolk lecithin, sodium oleate and sodium hydroxide), benzodiazepines, opioids, rocuronium bromide, sugammadex sodium and their drug components; those with cross-allergy to halogenated anesthetics, and those who had jaundice and unexplained high fever after using halogenated agents before are prohibited; those with contraindications for propofol.
* Having the following medical history or evidence that increases the risk of sedation/anesthesia collected before or during the screening:

  1. Cardiovascular history: uncontrolled hypertension or systolic blood pressure (SBP) > 160 mmHg and/or diastolic blood pressure (DBP) > 100 mmHg after treatment with antihypertensive drugs, severe arrhythmia, heart failure, Adams-stokes syndrome, unstable angina pectoris, myocardial infarction occurred within the recent 6 months before screening, a history of tachycardia/bradycardia requiring drug treatment, third-degree atrioventricular block.
  2. Respiratory history: respiratory insufficiency, a history of obstructive pulmonary disease, a history of bronchospasm requiring treatment within 3 months before screening, those who suffered from acute respiratory tract infection within 1 week before the baseline period and had one of the symptoms such as obvious fever, wheezing or expectorant cough.
  3. Neurological and psychiatric history: a history of craniocerebral injury, convulsions, epilepsy, intracranial hypertension, cerebral aneurysm, cerebrovascular accident; or a history of schizophrenia, mania, long-term use of psychotropic drugs, cognitive dysfunction, etc.
  4. Gastrointestinal history: a history of gastrointestinal retention, active bleeding, gastroesophageal reflux or obstruction, etc., and the investigator judges that it may lead to reflux aspiration.
  5. Diabetic patients with unsatisfactory blood glucose control (fasting blood glucose ≥ 11.1 mmol/L or random blood glucose ≥ 13.6 mmol/L).
  6. Having a history of diseases in the liver, kidney, blood system, nervous system or metabolic system that are not controlled and are judged by the investigator as not suitable for participating in this study and have significant clinical significance.
  7. A history of alcohol abuse within 3 months before screening.
  8. A history of drug abuse within 3 months before screening.
  9. Those who had severe infection, severe trauma or major surgical operations within 4 weeks before screening.
* Having any of the following risks in airway management before or during the screening:

  1. A history of asthma, wheezing.
  2. Those with sleep apnea syndrome.
  3. Those with a history or family history of malignant hyperthermia.
  4. Those with a history of failed tracheal intubation.
  5. The investigator judges that there is a difficult airway or it is determined as difficult tracheal intubation (modified Mallampati score is grade III or IV).
* Having used any of the following drugs or treatments before anesthesia induction:

  1. Those who participated in any drug clinical trials within 1 month before screening.
  2. Those who used propofol, other general sedative/anesthetic drugs and/or opioid analgesics or compound preparations containing opioid analgesic components within 4 hours before anesthesia induction.
* Laboratory examination indexes during the screening period meet the following standards and are confirmed by reexamination:

  1. Neutrophil count < 1.5 × 10⁹/L.
  2. Platelet count < 80 × 10⁹/L.
  3. Hemoglobin < 90 g/L (and without blood transfusion within 14 days).
* Pregnant and lactating women; fertile women or men who are unwilling to use contraception during the entire trial period; subjects (including male subjects) who have a pregnancy plan within 3 months after the trial.
* Subjects who are considered by the investigator to have any other factors that are not suitable for participating in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Optimize the parameters CeLoC/CeRoC and Ke0 of the target-controlled infusion model of cipepofol. | 2 h
  Calculate/record the effect-site concentrations of ciprofol (CeLoC/CeRoC) at the time of loss of consciousness (LoC) and recovery of consciousness (RoC), as well as the effect-site equilibrium rate constant (Ke0).
  The units of CeLoc and CeRoc is μg/ml. Calculate Ke0 through computer simulation based on the pharmacokinetic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Gao Jingui, Doctor, Principal Investigator — Investigator
Locations (2):
- China (2):
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No
Ce and Cp parameters